CLINICAL TRIAL: NCT03708510
Title: Clinical Evaluation of Two Low-shrinkage Composites After Different Preparation Techniques
Brief Title: Clinical Evaluation of Two Low-shrinkage Composites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Dr. Fatma Dilşad Öz, Doctor, DDS, PhD, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Kalore-Silorane, Laser-Bur
Record Dates: First submitted 2018-10-14; First posted 2018-10-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Tooth Diseases
MeSH Terms: conditions — Tooth Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Filtek Silorane-Er,Cr:YSGG Laser (Experimental)
  Interventions: Device: Restorative materials- Filtek Silorane; Device: Preparation-Er,Cr:YSGG Laser
- Filtek Silorane- Diamond Bur (Experimental)
  Interventions: Device: Restorative materials- Filtek Silorane; Device: Preparation- Diamond Bur
- Kalore- Er,Cr:YSGG Laser (Experimental)
  Interventions: Device: Restorative materials-Kalore; Device: Preparation-Er,Cr:YSGG Laser
- Kalore- Diamond Bur (Experimental)
  Interventions: Device: Restorative materials-Kalore; Device: Preparation- Diamond Bur

INTERVENTIONS:
Device: Restorative materials- Filtek Silorane — Filtek Silorane
  Arms: Filtek Silorane- Diamond Bur; Filtek Silorane-Er,Cr:YSGG Laser
Device: Restorative materials-Kalore — Kalore
  Arms: Kalore- Diamond Bur; Kalore- Er,Cr:YSGG Laser
Device: Preparation-Er,Cr:YSGG Laser — Er,Cr:YSGG Laser
  Arms: Filtek Silorane-Er,Cr:YSGG Laser; Kalore- Er,Cr:YSGG Laser
Device: Preparation- Diamond Bur — Bur
  Arms: Filtek Silorane- Diamond Bur; Kalore- Diamond Bur

SUMMARY:
Patients with 4 occlusal lesions in molar teeth will be included. Occlusal cavities will be prepared either by Er,Cr:YSGG laser (LS) or conventional diamond bur (BR). Cavities will be restored with Filtek Silorane (3M-ESPE) (SR) and with Kalore (GC) (KR) according to the manufacturers' instructions. All restorative procedures will be performed by one operator and the restorations will be examined by two evaluators according to the FDI (World Dental Federation) criteria at baseline and at 6-month, 1-, 2-,3-, 4-, 5-, 6-, 7-, 8-, 9-, 10-year. Patients' satisfaction about the preparation methods will be evaluated with a survey. Pearson Chi-Square test will be used for statistical analyze(p=0.05).

ELIGIBILITY:
Inclusion Criteria:

1. age range will be 18 to 60
2. patients should have at least 4 occlusal caries lesions require restoration
3. healty periodontal status
4. a good likelihood of recall availability

Exclusion Criteria:

1. poor gingival health
2. adverse medical history
3. potential behavioral problems

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-05-01 (Actual); Primary Completion 2011-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Clinical performance of different low-shrinkage composites and preparations | 10 years
  Evaluations according to FDI criteria